CLINICAL TRIAL: NCT04347148
Title: Postural and Clinical Outcomes of SNAGs Treatment in Cervicogenic Dizziness Patients: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniter Onlus (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Alessandro Micarelli, Scientific Director, Uniter Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniterSNAG
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Cervicogenic Dizziness; Rehabilitation
Keywords: cervicogenic dizziness; sustained natural apophyseal glides; posturography testing; fast Fourier transform; cervical range of motion

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated to SNAGs (n = 41) or placebo (n = 39) treatment, constituted by a detuned laser. Both groups received their interventions 6 times over 4 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNAGs treatment (Experimental): cervicogenic patients will undergo SNAGs treatment. Based on personal history, the offending active cervical movement (i.e. the movement predominantly causing dizziness) will be identified and treatment direction will be determined. As suggested, the active movement to most likely cause dizziness is cervical extension, though also rotation or flexion will be shown to provoke it. With the participant in an upright sitting position, a skilled physiotherapist (blinded to the allocation) will apply a sustained passive accessory movement (glide) while the participant will be asked to move actively as allowed by his/her physiological range in the direction producing their symptoms. This procedure will be repeated six times.
  Interventions: Procedure: SNAGs Treatment
- Detuned Laser (Placebo Comparator): cervicogenic patients will receive a sham treatment, carried out by the another skilled therapist (blinded to the allocation) and consisting in exposition to a detuned laser. A laser - deactivated by the manufacturer in order to produce no effective emission - will appear to operate normally, emitting a light signal and a beeping sound. Such procedure - which was shown to not activate somatosensory receptors and to have a very strong placebo effect - will be used for six applications, lasting 20 seconds, on various sites on the upper cervical spine, at a distance of 0.5-1cm from the skin.
  Interventions: Procedure: Sham Laser Treatment

INTERVENTIONS:
Procedure: SNAGs Treatment — a sustained passive accessory movement (glide), i.e. SNAGs, will be applied by the physiotherapist while the participant will be asked to move actively as allowed by his/her physiological range in the direction producing his symptoms.
  Arms: SNAGs treatment
Procedure: Sham Laser Treatment — A Laser YAG 3 Chronic (Winform Medical Engineering s.r.l., San Donà di Piave (VE), Italy), will be detuned and applied in the region of cervical spine in order to have a sham treatment
  Arms: Detuned Laser

SUMMARY:
Previous works demonstrated the relationship between postural disturbances and reduction in cervical range of motion (CROM) in patients suffering from cervicogenic dizziness (CGD). Since sustained natural apophyseal glides (SNAGs) have been proposed as an effective treatment, the aim of the present study was to evaluate how clinical measures could be affected in patients with cervicogenic dizziness undergoing SNAGs.

ELIGIBILITY:
Inclusion Criteria:

* accepted criteria will be operationalized to achieve the clinical suspicion of cervicogenic dizziness as following:

  1. Exclusion of these differential diagnoses: a. Migrainous vertigo b. Vertigo of central origin c. Benign paroxysmal positional vertigo (BPPV) d. Meniere disease e. Vestibular neuritis f. Vertigo induced by drugs g. Psychogenic vertigo (anxiety and/or panic disorder and/or phobia) h. Orthostatic hypotension
  2. presence of a subjective feeling of dizziness associated with pain, movement, rigidity, or certain positions of the neck at least from 3 months;
  3. Cervical pain, trauma, and/or disease
  4. If from traumatic origin, there has to be a temporal proximity between the onset of dizziness and the neck injury.

Diagnosis is positive if criteria 1 to 3 are fulfilled. As for criterion 2, dizziness had to occur during the same period than neck pain occurred and dizziness had to be proportional to the severity of the neck pain that generally fluctuates in time.

Criterion 4 addresses cervicogenic dizziness occurring after a neck trauma

Exclusion Criteria:

* presence of trauma or recent surgery in the head, face, neck, or chest;
* an otorhinolaryngological diagnosis of central or peripheral vertigo
* receiving physiotherapy during the study period.
* History, physical examination and a thorough clinical otoneurological examination will be devised to exclude extracervical causes of dizziness.
* In order to exclude vestibular hypofunction, video Head Impulse Test - and the technique proposed in previous studies will be used to study the vestibulo-ocular reflex.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Balance Test | one month
  Study of the surface of the ellipse of confidence (calculated in mm) by means of static posturography platform will be used to assess the sway of the posture. Low levels of outcomes indicate better performances. No specific reference ranges are given in literature.
Cervical Spine Movements | one month
  A cervical range of motion (CROM) goniometer, which has been shown to be a reliable tool with good validity, will be used to measure (in degrees) cervical spine movements. Active flexion, extension, left and right rotation, and left and right lateral flexion will be measured three times and then averaged. Low levels of outcomes indicate worse performances. No specific reference ranges are given in literature.

SECONDARY OUTCOMES:
Self-report dizziness | one month
  The Italian Dizziness Handicap Inventory (DHI) wil be used to assess the self-report dizziness handicap. It consists of 25 questions designed to assess a patient's functional (nine questions), emotional (nine questions), and physical (seven questions) limitations; absolute scores range from 0 to 100, with moderate and severe disability usually associated with scores above 30 and 60, respectively
Disability of the Neck | one month
  Level of neck spine disability will be assessed by means of Neck Disability Index (NDI). This self-report questionnaire has a single-factor structure comprising 10 items which assess different activities of daily living on a 6-point Likert-type scale (ranging from 0 to 5). Higher absolute scores indicate more severe pain and greater disability
Pain of the Neck | one month
  Neck Pain Intensity (NPI) will be evaluated with the visual analogue scale for pain. This self-report reliable tool consists of a 100-mm horizontal line between the extremes 'no pain' (left) and 'worst imaginable pain' (right).
Fear of Movement | one month
  Fear of movement will be quantified with the Tampa Scale for Kinesiophobia (TSK-17), a 17 item self-report questionnaire in which each question is scored using a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree); 4 items (4, 8, 12, and 16) are negatively worded and reverse scored. Higher absoute scores indicate a higher degree of kinesiophobia
Anxiety and Depression | one month
  Anxiety and depression will be evaluated with the Hospital Anxiety and Depression Scale (HADS). This self-administered questionnaire contains 14 items, rated on a 4-point Likert type scale (from 0 to 3 points). The tool includes 2 subscales of 7 items that assess anxiety and depression. Higher absolute scores indicate higher levels of anxiety and depression in the 2 subscales, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- UNITER ONLUS for balance and rehabilitation research, Guidonia, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hain TC. Cervicogenic causes of vertigo. Curr Opin Neurol. 2015 Feb;28(1):69-73. doi: 10.1097/WCO.0000000000000161. PMID 25502050
- [Result] Lystad RP, Bell G, Bonnevie-Svendsen M, Carter CV. Manual therapy with and without vestibular rehabilitation for cervicogenic dizziness: a systematic review. Chiropr Man Therap. 2011 Sep 18;19(1):21. doi: 10.1186/2045-709X-19-21. PMID 21923933
- [Result] Wrisley DM, Sparto PJ, Whitney SL, Furman JM. Cervicogenic dizziness: a review of diagnosis and treatment. J Orthop Sports Phys Ther. 2000 Dec;30(12):755-66. doi: 10.2519/jospt.2000.30.12.755. PMID 11153554
- [Result] Reid SA, Callister R, Katekar MG, Rivett DA. Effects of cervical spine manual therapy on range of motion, head repositioning, and balance in participants with cervicogenic dizziness: a randomized controlled trial. Arch Phys Med Rehabil. 2014 Sep;95(9):1603-12. doi: 10.1016/j.apmr.2014.04.009. Epub 2014 May 2. PMID 24792139
- [Result] Reid SA, Rivett DA, Katekar MG, Callister R. Sustained natural apophyseal glides (SNAGs) are an effective treatment for cervicogenic dizziness. Man Ther. 2008 Aug;13(4):357-66. doi: 10.1016/j.math.2007.03.006. Epub 2007 Oct 22. PMID 17951095
- [Result] Micarelli A, Viziano A, Augimeri I, Micarelli B, Capoccia D, Alessandrini M. Diagnostic route of cervicogenic dizziness: usefulness of posturography, objective and subjective testing implementation and their correlation. Disabil Rehabil. 2021 Jun;43(12):1730-1737. doi: 10.1080/09638288.2019.1680747. Epub 2019 Oct 26. PMID 31656108
- [Result] Grande-Alonso M, Moral Saiz B, Minguez Zuazo A, Lerma Lara S, La Touche R. Biobehavioural analysis of the vestibular system and posture control in patients with cervicogenic dizziness. A cross-sectional study. Neurologia (Engl Ed). 2018 Mar;33(2):98-106. doi: 10.1016/j.nrl.2016.06.002. Epub 2016 Jul 21. English, Spanish. PMID 27452617